CLINICAL TRIAL: NCT06816446
Title: Testing the Efficacy of Rodenstock Spectacle Lenses in Myopia Progression: a Two Year Clinical Trial
Brief Title: Influence of Rodenstock Spectacle Lenses on Myopia Progression.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rodenstock GmbH (Industry)
Collaborators: National University of Singapore (Other); National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Chen-Hsin Sun, Dr. Sun Chen-Hsin; Dr. Raymond Najjar, Rodenstock GmbH
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CTS01245
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Myopia
Keywords: Myopia; Myopia control; Lenses; Light
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Myopia control spectacle lens
  Interventions: Device: Myopia control spectacle lens
- Control group (Active Comparator): Single-vision spectacle lens
  Interventions: Device: Single-vision lens

INTERVENTIONS:
Device: Myopia control spectacle lens — The intervention group will wear specially designed lenses that aim to slow the progression of myopia. Follow-up visits will take place at regular intervals.
  Arms: Intervention group
Device: Single-vision lens — The control group will wear single vision lenses for one year. They will then switch to the myopia control lens for a further year. Follow-up visits will take place at regular intervals.
  Arms: Control group

SUMMARY:
The prevalence of myopia in Singapore is among the highest in the world, with 65 percent of our children being myopic by Primary 6, and 83 percent of young adults being myopic. As such, Singapore is often labelled as the "Myopia Capital of the World". By 2050, it is projected that 80 to 90 per cent of all Singaporean adults above 18 years old will be myopic and 15 to 25 percent of these individuals may have high myopia.

High myopia (spherical equivalent refraction ≤ -5 D) puts one at risk of many eye disorders later in life, such as early cataracts, glaucoma and macular degeneration. These complications often cause significant morbidity and may even be sight-threatening. Hence there is an urgent and growing need for synergistic efforts to counter myopia.

The goal of this clinical trial is to test the efficacy of spectacle lenses in controlling the progression of myopia in children (aged 6-12 years) over a period of 2 years. In addition, this trial aims to evaluate the impact of these spectacle lenses on central visual performance and visual comfort.

Therefore, in this randomised, double-masked clinical trial, one hundred and eighty-five (n=185) subjects aged 6-12 years with mild or moderate myopia (< -5D) will be randomised in a 1:1 allocation ratio into three strata defined by age 6-8, 8-10 and 10-12 years to ensure age balance between the two arms (control group - single vision lenses and intervention group - myopia control lenses, gender matched). In the control group, after one year (12 months) of wearing single vision lenses, the children will switch to the myopia control lenses (crossover design).

ELIGIBILITY:
Inclusion Criteria:

* All myopic children aged 6-12 years old
* Treatment naïve
* Sphere: -0.5 D till -5.00 D
* Anisometropia < 1.5D
* Astigmatism > -1.5D
* Monocular best corrected visual acuity +0.1 logMAR or better, and binocular visual acuity 0.0 logMAR or better

Exclusion Criteria:

* On current myopia control treatments
* Any diagnosed ocular conditions besides myopia or astigmatism.
* No diagnosed ocularmotor conditions (Nystagmus, strabismus, etc.)
* Any diagnosed chronic physical or mental disabilities
* Contraindication in cycloplegia (high IOP, etc.)
* Corneal astigmatism > 1.5 D; irregular astigmatism

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 185 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Spherical equivalent refraction | 2 years
  Change in spherical equivalent refraction

SECONDARY OUTCOMES:
Axial length | 2 years
  Change in axial length from baseline
Peripheral refraction | 2 years
  Change in peripheral refraction from baseline
Choroidal thickness | 2 years
  Change of choroidal thickness from baseline
Visual acuity | 1 year
  Difference in central visual acuity between single vision lenses and myopia control lenses
Contrast sensitivity | 1 year
  Difference in contrast sensitivity between single vision lenses and myopia control lenses
Visual comfort | 1 year
  Difference in visual comfort between single vision lenses and myopia control lenses
Light exposure | 2 years
  Impact of light exposure characteristics on myopia progression

CONTACTS AND LOCATIONS:
Locations (1):
- NUH, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Team is undecided whether to share or not share the data. This may be amended.